CLINICAL TRIAL: NCT03617016
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Prospective Pilot Study to Preliminarily Evaluate the Efficacy of Domperidone in Adult Chinese Subjects With Functional Dyspepsia
Brief Title: Preliminarily Evaluate the Efficacy of Domperidone in Adult Chinese Participants With Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108512; R033812DYP4002 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2018-07-10; First posted 2018-08-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Domperidone (Experimental): Participants will receive domperidone 10 milligram (mg) tablets orally thrice in a day from Day 1 to Day 14.
  Interventions: Drug: Domperidone
- Placebo (Placebo Comparator): Participants will receive matching placebo corresponding to domperidone orally thrice in a day from Day 1 to Day 14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Domperidone — Participants will receive domperidone tablets orally.
  Other Names: JNJ-17296812
  Arms: Domperidone
Drug: Placebo — Participants will receive matching placebo to domperidone tablets orally.
  Arms: Placebo

SUMMARY:
The main purpose of the study is to assess the efficacy of domperidone in treatment of functional dyspepsia (FD) in Chinese participants and identify sub-populations (subtype of the disease) who are sensitive to domperidone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the diagnostic criteria for functional dyspepsia (Postprandial Distress Syndrome [PDS] and/or Epigastric Pain Syndrome [EPS]) according to Rome IV diagnostic criteria for functional gastrointestinal disorders before and through screening
* Must have had an upper endoscopy that shows no evidence of structural change that is likely to explain the dyspepsia symptoms. If the participant has had the upper endoscopy performed within 3 months before screening, no re-test is needed
* Must have an abdominal ultrasonography that shows no evidence of organic disease that is likely to explain the dyspepsia symptoms. If the participant has the abdominal ultrasonography performed within 3 months before screening, no re-test is needed
* A woman of childbearing potential must have a negative serum (beta human chorionic gonadotropin [beta-hCG]) pregnancy test at Screening
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 30 days after receiving the last dose of study drug
* Otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and signed by the investigator. Specifically, for vital signs, the participant must have blood pressure (after participant has been supine for 10 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic (inclusive) and between 60 and 90 mmHg diastolic (inclusive)

Exclusion Criteria:

* Has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease (including bronchospastic respiratory disease), diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Has history of risk factors for Torsade de Pointes or family history of short QT syndrome, long QT syndrome, sudden unexplained death at a young age (less than or equal to [<=] 40 years); or a history of second- or third-degree heart block
* Has clinically significant electrolyte disorders or conditions that result in electrolyte disorders, such as severe dehydration, vomiting, malnutrition, eating disorders, renal diseases, or the use of potassium-wasting diuretics or insulin in acute settings
* Has a history of esophageal, gastric, or duodenal surgery, including endoscopic surgery
* Has any condition in which stimulation of gastric motility might be dangerous, for example (e.g.), in the presence of gastrointestinal (GI) hemorrhage, mechanical obstruction, or perforation
* Has used any of the following medications 7 days before screening: proton pump inhibitors, antacids, anti-secretory agents, histamine2 receptor antagonists, gastric mucosa protective agents, digestive enzymes, prokinetic agents (including macrolide antibiotics), and other drugs that affect gastrointestinal function, QT-prolonging drugs, cytochrome P450 3A4 inhibitors, monoamine oxidase inhibitors (MAOIs), nonsteroidal anti-inflammatory agents, aspirin (including low-dose aspirin), anticholinergics, antidepressants, or diuretics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Response Rate Based on Overall Treatment Effect (OTE) | Day 14
  Participants with overall symptoms extremely improved or improved will be considered as responders. Response rate of OTE is defined as the percentage (%) of responders in total participants.

SECONDARY OUTCOMES:
Response Rate Based on OTE | Day 7
  Participants with overall symptoms extremely improved or improved will be considered as responders. Response rate of OTE is defined as the percentage of responders in total participants.
Percentage of Participants with Each Average Symptom Score Decreased at least 2 Points Compared to Baseline | Baseline, Day 1 to Day 7 and Day 8 to Day 14
  Participants on every need will rate the severity of functional dyspepsia (FD) symptoms (postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea and vomiting) on a Likert scale of 7-point using e-diaries, the score range is 1 to 7. The higher the score, the more serious the outcome is.. For each FD symptom, the percentage of participants with each average symptom score (average of Day 1 through Day 7 and Day 8 through Day 14) decreased at least 2 points compared to baseline will be calculated.
Change From Baseline in Frequency of Each FD Symptom | Baseline to Day 7 and Day 15
  Participants on every need will rate the severity of functional dyspepsia (FD) symptoms (postprandial fullness, early satiation, epigastric pain, epigastric burning, belching, epigastric bloating, nausea and vomiting) on a Likert scale of 7-point using e-diaries, the score range is 1 to 7. The higher the score, the more serious the outcome is.
Change from Baseline in Disease-Speciﬁc Quality of Life (QoL) in FD as Assessed by Nepean Dyspepsia Index (NDI) Score | Baseline and Day 15
  QoL will be assessed by using the NDI questionnaire. The NDI is a reliable and valid measure of quality of life in FD. The NDI originally contains 42 items designed to measure impairment of a subjective ability engaged in relevant aspects of their life because of dyspepsia. The score range is 0 to 100. The higher the score, the more serious the outcome is.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (5):
- China (5):
  - Capital Medical University, Beijing Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Fujian Provincial Hospital, Fuzhou
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan

REFERENCES:
- See also: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Prospective Pilot Study to Preliminarily Evaluate the Efficacy of Domperidone in Adult Chinese Subjects with Functional Dyspepsia — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108512&attachmentIdentifier=9a064ba5-877b-49b8-9721-0f22d04b22ea&fileName=CR108512_CSR_Synopsis.pdf&versionIdentifier=